CLINICAL TRIAL: NCT02400216
Title: A Multidisciplinary Approach to Deciphering the Mechanisms Involved In Microbial Translocation Across the Spectrum of HCV Associated Liver Fibrosis
Brief Title: Deciphering the Mechanisms Involved in Microbial Translocation Across the Spectrum of HCV Associated Liver Fibrosis
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150100; 15-DK-0100
Record Dates: First submitted 2015-03-26; First posted 2015-03-27 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-04-09

CONDITIONS: Cirrhosis
Keywords: Chronic Hepatitis C; Cirrhosis; Liver Biopsy; Microbiome; Natural History
MeSH Terms: conditions — Fibrosis; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients with fibrosis levels spanning from bridging fibrosis to cirrhosis (Ishak fibrosis score 5-6)
  Interventions: Drug: dual cholate
- Group B: Patients with minimal fibrosis (Ishak score 0-1).
  Interventions: Drug: dual cholate

INTERVENTIONS:
Drug: dual cholate — test for defining disease severity

SUMMARY:
Background:

- Hepatitis C infection (HCV) is a leading cause of liver disease. Normal bacteria from the intestines may spread to the liver and blood during liver disease. This is called bacterial translocation (BT). Researchers think BT may cause liver disease to worsen.

Objectives:

- To study the mechanisms involved in BT in early and advanced liver disease. To find out whether BT causes liver disease to worsen.

Eligibility:

- People over age 18 with HCV and clinically stable liver disease.

Design:

* Participants will be screened with medical history and physical exam. They will have blood tests and imaging studies.
* Participants will have 2 outpatient visits and a 3-day stay at the clinic.
* At visit 1, participants will have urine and blood tests. They will have a magnetic resonance imaging (MRI) scan. A solution will be injected into a vein. The MRI scanner is a metal cylinder surrounded by a magnetic field. The participant will lie on a table that slides in and out of the cylinder.
* At visit 2, a substance will be injected into a vein and swallowed. Participants will then have blood drawn 5 times over 90 minutes.
* During the inpatient stay, serial blood tests will be drawn.
* Participants will give 2 stool samples and have another MRI.
* A needle will be inserted through the chest wall into a vein inside the liver, guided by ultrasound. The blood pressure inside this vein will be measured and blood will be drawn from it. About 1 inch of liver tissue will be removed.
* A study investigator will call participants to discuss all test results.

DETAILED DESCRIPTION:
Hepatitis C (HCV) is a leading cause of cirrhosis worldwide. Most complications associated with cirrhosis are driven by an altered portal circulation and the development of portal hypertension. Bacterial translocation (BT) from the gut to the systemic circulation is considered a pivotal mechanism contributing to the development of life-threatening complications in end stage cirrhosis. Recent evidence suggests that the liver and systemic circulation may be exposed to gut derived microbial products at earlier stages of liver disease. This early exposure may trigger hepatic inflammation, modify immune host response and accelerate hepatic fibrogenesis; which, in turn, impairs portal inflow, alters the portal circulation, and leads to development of portal hypertension. The mechanisms resulting in systemic exposure to gut derived microbial products, and the subsequent host response to BT has not been studied in patients with early liver disease nor fully compensated cirrhosis.

We therefore intend to enroll 30 chronic HCV patients with either cirrhosis (20) or minimal liver fibrosis (10). Study participants will undergo extensive evaluation with portal vein sampling and pressure measurements, dual cholate clearances, liver biopsy, serologic, immunologic, fecal microbiome and imaging studies. This will be followed by an optional second percutaneous liver biopsy and portal vein sampling 9-15 months after HCV treatment. The treatment protocol is a separate independent protocol, 15-DK- 0143 utilizing Sofosbuvir and GS-5816. The goals of our study are to characterize the extent of BT in early stages of cirrhotic and non-cirrhotic liver disease, explore the mechanisms contributing to its occurrence and identify potential serological, immunological and hemodynamic biomarkers associated with chronic infection. This, in turn, can aid in establishing a possible link between BT, subsequent host responses and severity of liver disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. All age greater than 18 male or female
  2. Capacity to provide written informed consent
  3. Evidence of HCV RNA in 2 serum samples at least 6 months apart.
  4. All HCV genotypes
  5. Liver biopsy in the last 2 years prior to enrollment showing Ishak fibrosis score of either 0-1 or 5-6. An alternative to liver biopsy will be a Fibroscan study performed in the 6 months prior to study enrollment showing a score of either kPa <7 or above 13.
  6. Child-Pugh score less than or equal to 6
  7. Prior to each liver biopsy and portal vein cannulation procedure, blood will be drawn for CBC, PT/INR & acute care panel.

EXCLUSION CRITERIA:

1. Pregnant women or females at child bearing age not taking measures to prevent pregnancy during the period of study
2. Patients currently on treatment for hepatitis C
3. Clinical, serologic or histopathologic evidence supporting other etiologies of chronic liver disease besides HCV
4. Current or past clinical evidence of decompensated liver disease (e.g. ascites, bleeding esophageal varices, spontaneous bacterial peritonitis, encephalopathy etc.)
5. Cross sectional liver imaging study from the past 6 months showing a focal lesion suspicious of hepatocellular carcinoma and/or alpha-fetoprotein level greater than 200 ng/mL.
6. Patients with active bacterial, viral or fungal, systemic or localized infection.
7. Antibiotic treatment 30 days prior to study enrollment
8. History of chronic inflammatory diseases of the bowel (Crohn s disease, Ulcerative colitis and celiac disease)
9. History of congestive heart failure of moderate to severe degree.
10. History of non-cirrhotic portal hypertension or portal vein thrombosis
11. Patients with severe allergic reactions to iodine contrast, which cannot be controlled by premedication with antihistamines and steroids.
12. EXCLUSION CRITERIA FOR MRI:

    12.1 Subjects with contraindication to MRI scanning. These contraindications include but are not limited to the following devices or conditions:

    <TAB>a. Implanted cardiac pacemaker or defibrillator

    <TAB>b. Cochlear Implants

    <TAB>c. Ocular foreign body (e.g. metal shavings)

    <TAB>d. Embedded shrapnel fragments

    <TAB>e. Central nervous system aneurysm clips

    <TAB>f. Implanted neural stimulator

    <TAB>g. Medical infusion pumps

    <TAB>h. Any implanted device that is incompatible with MRI.

    12.2 Unsatisfactory performance status as judged by the referring physician such that the subject could not tolerate an MRI scan. Examples of medical conditions that would not be accepted would include unstable angina and dyspnea at rest.

    12.3 Subjects requiring sedation for MRI studies.

    12.4 Subjects with a condition precluding entry into the scanner (e.g. morbid obesity, claustrophobia, etc.).

    12.5 Pregnant or lactating women.

    12.6 Subjects with severe back-pain or motion disorders who will be unable to tolerate supine positioning within the MRI scanner and hold still for the duration of the examination.

    12.7 For Gadolinium based and SPIO MRI Use:

    <TAB>a. History of severe allergic reaction to these contrast agents despite the use of premeditation with an anti-histaminic and cortisone.

    <TAB>b. eGFR < 60 ml/min/1.73m^2
13. Absolute neutrophil count below 1000/mm^3, Hemoglobin level below 10.0 g/dl or platelet count lower than 70,000/mm^3.
14. INR greater than or equal to 1.5, PTT greater than or equal to 1.3 times control and/or any known history of disease associated with increased bleeding diathesis.
15. Serum creatinine greater than or equal to 2.0 mg/dl unless the measured creatinine clearance is greater than 60 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical patients with chronic HCV infection divided into 2 groups according to liver fibrosis stage.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Microbial product detection rate | Before anti viral therapy and 9-15 months after treatment
  Assess the extent of BT, explore possible mechanisms accounting for its occurrence and evaluate its effects on the immune system in different stages of liver fibrosis

SECONDARY OUTCOMES:
Dual-cholate liver function tests | Baseline, and 9-15 months after treatment
  Comparison of dual-cholate liver function tests and its association with microbial product levels in portal and systemic blood, between group A and group B patients.
SPIO-MRI Kupffer cell uptake | Baseline, and 9-15 months after treatment
  Comparison of SPIO-MRI Kupffer cell uptake values and its association with microbial product levels in portal and systemic blood between group A and group B patients.
Immune activation markers | Baseline, and 9-15 months after treatment
  Comparison of immune activation markers to bacterial products in liver tissue between group A and group B patients before and after HCV treatment.
Pro and anti-inflammatory gene transcription | Baseline, and 9-15 months after treatment
  Comparison of pro and anti-inflammatory gene transcription analysis in between group A and group B patients
Fecal microbiome | Baseline, and 9-15 months after treatment
  Comparison of fecal microbiome analysis between group A and group B patients
Species homology | Baseline, and 9-15 months after treatment
  Evaluation of species homology between microbial DNA identified in portal and systemic blood and fecal samples by deep sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-DK-0100.html